CLINICAL TRIAL: NCT04060654
Title: An Open-label, Treatment Extension Study for the Rapid Initiation of Extended-Release Buprenorphine Subcutaneous Injection (SUBLOCADE™)
Brief Title: SUBLOCADE Rapid Initiation Extension Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDV-6000-404
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder, Severe; Opioid Use Disorder, Moderate
MeSH Terms: conditions — Opioid-Related Disorders; Lymphoma, Follicular | interventions — Sublocade

STUDY DESIGN:
Intervention Model Description: After an initial injection of 300mg SUBLOCADE, all subjects will receive SUBLOCADE doses of 100mg or 300mg based on the medical judgement of the Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SUBLOCADE (Experimental): All subjects will receive SUBLOCADE 300mg on Day 1, followed by injections every 4 weeks at a dose determined by the Investigator (either 100 mg or 300 mg) for up to 5 total injections
  Interventions: Drug: Sublocade

INTERVENTIONS:
Drug: Sublocade — SUBLOCADE to be administered approximately every 4 weeks per local standard of care
  Other Names: Extended release buprenorphine

SUMMARY:
A single center, open-label SUBLOCADE treatment extension study in which up to 25 participants diagnosed with moderate to severe opioid use disorder (OUD) could be enrolled.

DETAILED DESCRIPTION:
This study is being conducted to assess the longer-term safety of an abbreviated initiation protocol of SUBLOCADE in subjects who have completed the INDV-6000-403 study. It is also to provide treatment to these individuals while they seek longer-term treatment arrangements, as on average it can take an individual with opioid use disorder (OUD) 6 months between seeking treatment and achieving an appointment at a provider in the United States (US).

Subjects who have completed the end of treatment (EOT) procedures for the INDV-6000-403 study may be eligible for participation. It is planned that the EOT visit for INDV-6000-403, which will occur approximately 28 days after the subject's first dose of SUBLOCADE, and Day 1 for INDV-6000-404 will occur within 2 days of the EOT visit, and that EOT assessments will serve as the screening assessments for this study.

On Day 1, eligible subjects will receive a subcutaneous (SC) injection of 300 mg SUBLOCADE. Subjects will return to the clinic for subsequent injections approximately every 4 weeks for a total of up to 5 injections. Adverse events and concomitant medications will be captured throughout the study, female subjects of childbearing potential will receive urine pregnancy tests and all subjects will have urine drug screening (UDS) and evaluation of the previous injection site performed. Subjects will otherwise be treated in accordance with local standard of care, and SUBLOCADE doses will be based on the medical judgment of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF) and have the ability to comply with the requirements and restrictions listed therein.
* Completed the EOT Visit for the INDV-6000-403 Study.
* Is an appropriate candidate in the opinion of the Investigator or medically qualified sub-Investigator.

Exclusion Criteria:

* Subject compliance issues during participation in the INDV-6000-403 study which, in the opinion of the Investigator, could potentially compromise subject safety.
* Subjects who are unable, in the opinion of the Investigator or Indivior, to comply fully with the study requirements including those who are currently incarcerated or pending incarceration legal action.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hassman, Principal Investigator — Hassman Research Institute
Locations (1):
- Hassman Research Institute, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mariani JJ, Dobbins RL, Heath A, Gray F, Hassman H. Open-label investigation of rapid initiation of extended-release buprenorphine in patients using fentanyl and fentanyl analogs. Am J Addict. 2024 Jan;33(1):8-14. doi: 10.1111/ajad.13484. Epub 2023 Nov 8. PMID 37936553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 participants who completed the INDV-6000-403 study were screened and enrolled into this extension study.
Groups:
- SUBLOCADE: All subjects will receive SUBLOCADE 300mg on Day 1, followed by injections every 4 weeks at a dose determined by the Investigator for up to 5 total injections
  Sublocade: SUBLOCADE to be administered approximately every 4 weeks per local standard of care
Period: Overall Study
Arm/Group | SUBLOCADE
Started | 17
Completed | 11
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- SUBLOCADE: All subjects will receive SUBLOCADE 300mg on Day 1, followed by injections every 4 weeks at a dose determined by the Investigator (either 100mg or 300mg) for up to 5 total injections
  Sublocade: SUBLOCADE to be administered approximately every 4 weeks per local standard of care
Arm/Group | SUBLOCADE
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (12.68)
Age, Customized [Count of Participants; unit: Participants]
  ≥18 to <30 | 4
  ≥30 to <45 | 6
  ≥45 to <60 | 5
  ≥60 to ≤ 65 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 5
  White | 10
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Screening body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.81 (4.181)
Screening BMI Group [Count of Participants; unit: Participants]
  0 to <18.5 (Underweight) | 2
  ≥18.5 and <25 (Normal) | 12
  ≥25 and <30 (Overweight) | 1
  ≥30 (Obesity) | 2
Tobacco Use [Count of Participants; unit: Participants]
  Never | 2
  Current | 15
Caffeine Use [Count of Participants; unit: Participants]
  Never | 2
  Current | 15
Opioids - Lifetime Use [Mean (Standard Deviation); unit: years] | 16.16 (15.246)
Opioids - Last 30 Days Prior to INDV-6000-403 Screening Visit [Mean (Standard Deviation); unit: Days] | 29.29 (2.910)
Opioids - Use via Intravenous Route in Last 30 Days [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Event (TEAE) Occurrence
Description: Study will report the number of participants with the occurrence of any TEAE during the treatment period.
Time Frame: From time of informed consent at Day 1 until EOT, assessed up until Day 141
Population: The safety population was used for the safety analysis, and consisted of all participants who received at least 1 dose of SUBLOCADE
Measure: Count of Participants; unit: Participants
Groups:
- SUBLOCADE: Participants who completed the INDV-6000-403 study and met study inclusion and exclusion criteria were given the option to enroll in this study. Baseline measures from the INDV-6000-403 study served also as baseline measures for this study. A total of 17 participants were screened and a total of 17 (100%) were enrolled into the study and received SUBLOCADE 300 mg at injection 1; subsequent doses could be reduced to 100 mg at the discretion of the investigator. Participants returned to the clinic approximately every 4 weeks for injection site assessments, urinary drug screens, pregnancy tests if applicable, subsequent injections and were assessed for the occurrence of any TEAEs. All other interventions were per clinic standard of care.
Arm/Group | SUBLOCADE
Number analyzed (Participants) | 17
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study Day 1 through end of treatment (EOT), up to Day 141
Groups:
- SUBLOCADE: All subjects will receive SUBLOCADE 300mg on Day 1, followed by injections every 4 weeks at a dose determined by the Investigator (either 100mg or 300 mg) for up to 5 total injections
  Sublocade: SUBLOCADE to be administered approximately every 4 weeks per local standard of care
Arm/Group | SUBLOCADE
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
The goal of the study was to assess the longer term safety of an abbreviated initiation protocol of SUBLOCADE and to provide treatment to these individuals while they seek longer term care arrangements. The COVID-19 pandemic, which began during the study period, potentially affected participant's ability to attend clinic visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will not disseminate, present or publish any of the study data without the prior written approval from Indivior to do so.

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04060654/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT04060654/SAP_000.pdf